CLINICAL TRIAL: NCT05830617
Title: Assessment and Modulation of Cortical Gamma Synchrony to Predict and Improve Stroke Recovery
Brief Title: Modulation of Cortical Gamma Synchrony in Stroke
Acronym: GAMMASTROKE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.08
Record Dates: First submitted 2023-03-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: tACS; gamma synchrony
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental): Real tACS will be delivered by applying two conductive electrodes over the left and right central areas, for 30 minutes/day (Monday-to-Friday), for two weeks, with the following parameters: sinewaves at 40Hz, peak-to-peak amplitude=1mA, 3s ramping-up and ramping-down. Intensity will be lowered if perceived as uncomfortable.
  Interventions: Device: real tACS
- sham tACS (Sham Comparator): Sham tACS will consist of only 30s of stimulation.
  Interventions: Device: sham tACS

INTERVENTIONS:
Device: real tACS — The effect of transcranial alternating current stimulation (tACS) will be investigated in WP3. Patients will undergo standard intensive rehabilitation plus gamma tACS for two weeks.
  Arms: real tACS
Device: sham tACS — In WP3, patients will undergo standard intensive rehabilitation plus sham tACS for two weeks.
  Arms: sham tACS

SUMMARY:
In the last decades, the research in neuroimaging-informed stroke prognosis and treatment has had a little clinical impact, often because of the costs of bringing complex procedures to the bedside. Cerebral stroke remains the leading cause of disability, with 65% of survivors chronically impaired at 6 months. Gamma synchrony (GS) is a fundamental mechanism of cortical function and can be estimated and modulated in a simple, inexpensive, and reliable way. It has provided valuable and cost-effective guidance in several neuropsychiatric conditions. In previous studies, we developed simple yet robust methods for assessing and manipulating GS and proved its relationship with clinical impairment in preliminary data.

The aim of the present project is to predict and improve stroke recovery by leveraging cortical mapping and modulation of GS via transcranial alternating current stimulation (tACS), a safe and inexpensive technique. The project capitalizes on technology readily available to the Italian national health system.

DETAILED DESCRIPTION:
The project will consist of 3 Work Packages (WPs):

* The aim of WP1 is to map the relationship between GS and clinical outcomes with EEG.
* The aim of WP2 is to translate GS assessment and modulation to bedside.
* The aim of WP3 is to modulate GS to improve rehabilitation outcomes.

ELIGIBILITY:
The participants in this study will be 140 stroke patients rehabilitated at IRCCS San Camillo hospital. 80 will participate in the WP1 and the WP2, while 60 will participate in the WP3 study. In WP1, data will also be collected on 80 healthy volunteer participants, approximately the same age as the patients.

Inclusion Criteria (healthy participants)

- no neurological or psychiatric disorder

Inclusion Criteria (patients)

* right or left hemisphere damage
* unilateral stroke
* no comorbidities with psychiatric disorders

Exclusion Criteria (general):

* Diagnosis of epilepsy or family history up to the second degree with it
* Episodes of febrile convulsions or recurrent fainting
* Head trauma
* Presence of surgical clips or metal implants in the head
* Diagnosis of heart disease
* Presence of a cardiac pacemaker or artificial heart valve
* Presence of hearing aids/prostheses
* Hearing problems or tinnitus
* Vision problems not corrected with lenses (such as color blindness)
* Taking tricyclic antidepressant medications
* Taking neuroleptic medications
* Diagnosis of headache or migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-03-23 (Estimated); Study Completion 2024-03-23 (Estimated)

PRIMARY OUTCOMES:
Gamma synchrony Work Package 1 (WP1) | baseline
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Gamma synchrony Work Package 1 (WP1) | immediately after the intervention
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Gamma synchrony Work Package 3 (WP3) | baseline
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Gamma synchrony Work Package 3 (WP3) | immediately after the intervention
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Gamma synchrony (reduced number of EEG sensors). Work Package 2 (WP2) | baseline
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Gamma synchrony (reduced number of EEG sensors). Work Package 2 (WP2) | immediately after the intervention
  Gamma synchrony will be measured via exposure to amplitude-modulated 40Hz sounds (5 min, sequence of amplitude-modulated tones at 40 Hz, delivered via earplug binaurally). Gamma synchrony will be quantified as power of the EEG gamma band. Gamma synchrony will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)

SECONDARY OUTCOMES:
Behavioral performance (response times). Work Package 1 (WP1) | baseline
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of response times (how fast the participants complete the task). Behavioral performance will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (response times). Work Package 1 (WP1) | immediately after the intervention
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of response times (how fast the participants complete the task). Behavioral performance will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (response times). Work Package 3 (WP3) | baseline
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of response times (how fast the participants complete the task). Behavioral performance will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (response times). Work Package 3 (WP3) | immediately after the intervention
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of response times (how fast the participants complete the task). Behavioral performance will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (accuracy). Work Package 1 (WP1) | baseline
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of accuracy (% of correct responses). Behavioral performance will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (accuracy). Work Package 1 (WP1) | immediately after the intervention
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of accuracy (% of correct responses). Behavioral performance will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (accuracy). Work Package 3 (WP3) | baseline
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of accuracy (% of correct responses). Behavioral performance will be measured at the baseline of the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)
Behavioral performance (accuracy). Work Package 3 (WP3) | immediately after the intervention
  Participants' cognitive performance at neuropsychological tests will be measured. Behavioral performance will be measured in terms of accuracy (% of correct responses). Behavioral performance will be measured immediately after the intervention (i.e., standard intensive rehabilitation at IRCCS S. Camillo Hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Arcara, Principal Investigator — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice, Italy

IPD SHARING:
Plan to Share IPD: No